CLINICAL TRIAL: NCT04100239
Title: A Pilot and Feasibility Trial of a Group Mindfulness and Self-compassion Intervention for Young People Diagnosed With Inflammatory Bowel Disease
Brief Title: A Pilot and Feasibility Trial of a Group Mindfulness and Self-compassion Intervention for Young People Diagnosed With IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 159047
Record Dates: First submitted 2019-09-05; First posted 2019-09-24 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel disease; mindfulness; self-compassion; young people; pilot study
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: This study is designed as a pilot and feasibility trial, using a stepwedged design. Pilot trials are used in advance of a larger future definitive randomised controlled trial (RCT) to focus on the development and refinement of the intervention, assess potential effectiveness, intervention acceptability and to determine whether a larger RCT is feasible. In step-wedged designs, all participants begin the study as 'control participants' and at regular 'steps' one group is crosses from the control to the intervention condition, until all groups have completed the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Open continuous recruitment of participants to trial where all participants begin the study as 'control participants' and at regular 'steps' participants are allocated to next available intervention group and cross from the control to the intervention condition, until all groups have completed the intervention.
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — MBSR is designed to complement any existing medical treatments, and focuses on the development of mindfulness meditation practice to alleviate psychological distress. MBCL is designed as a follow-up intervention to MBSR and aims to help individuals to turn towards suffering and developing a kind attitude to the self.
  Other Names: Mindfulness-based compassionate living (MBCL)

SUMMARY:
Young people with IBD face all the usual complexities of growing up, with the additional complications of having a chronic health condition, often recently diagnosed, which can have a detrimental impact on their mental health.

This research seeks to examine the potential effectiveness of a two-stage intervention for young people with IBD via a pilot feasibility trial. First, a mindfulness-based stress reduction (MBSR) group with a "Mindfulness based compassionate living" (MBCL) group delivered soon afterwards. Both interventions will be delivered online. MBSR aims to increase peoples awareness of their tendency to get caught up in thoughts and help them live in the present moment. Once an individual has achieved greater awareness of their thought processes, MBCL then aims to help individuals to become kinder to themselves, and less critical. We know from interview studies with young people with IBD that they can be harsh on themselves about how they are coping, and being harsh and critical can impact wellbeing. By targeting mindfulness and self-compassion we hope to demonstrate a positive impact on wellbeing, by reducing stress, anxiety and depression and improving quality of life (primary outcome measures) for young people with IBD and equip them with a mindfulness practice to use in the future as they continue to manage their IBD.

DETAILED DESCRIPTION:
Design: This study is designed as a pilot and feasibility trial, using a step-wedged design, and designed in line with CONSORT guidance. Pilot trials are used in advance of a larger future definitive randomised controlled trial (RCT) to focus on the development and refinement of the intervention, assess potential effectiveness, intervention acceptability and to determine whether a larger RCT is feasible. In step-wedged designs, all participants begin the study as 'control participants' and at regular 'steps' one group crosses from the control to the intervention condition, until all groups have completed the intervention. The step-wedged design is a pragmatic and financially viable design which reconciles the need for robust evaluations and logistical time constraints, as each participant acts as their own control. On conclusion of group participation, all participants will be invited to take part in one-to-one interviews with the lead researcher to discuss their experiences of MBSR+MBCL, to assess the acceptability of the intervention and inform future adaptations prior to larger trial.

Recruitment: Eligible and consenting participants will be identified in two ways. Firstly, by clinical staff at either Sheffield Teaching Hospital (NHS) or Sheffield Children's Hospital specialist IBD gastroenterology services and secondly, by poster, email or social media advertisements at the University of Sheffield and through relevant charitable organisations. Participants will be recruited on an ongoing basis and allocated to the next available group, or another, if the dates of the next group are not convenient.

Procedure: All consenting and eligible participants will meet with the lead researcher who will induct them into the trial and inform them of group allocation, and when they will commence the intervention. As in most psychological intervention trials, it will be impossible to blind participants to the interventions they are receiving. All outcome measures will be completed online via the Qualtrics platform.

Interventions (delivered online via video call): MBSR is an 8-week intervention consisting of 2.5 hour weekly sessions which involves the teaching and practice of formal mindfulness exercises, aimed at promoting the use of mindfulness in daily life for individuals experiencing stress, pain and/or illness. Participants are asked to engage in homework exercises which are intended to reinforce the techniques learnt each week. The intervention will aim to establish home practice and introduce self-compassion. MBCL is designed to be a follow-up intervention to a MBI. MBCL is a group intervention, also eight weeks in length and the sessions last 2.5 hours. The sessions contain a mixture of mindfulness practice, group discussion and didactic and interactive teaching. However, the content of the practices are different to traditional MBSR, focusing on turning towards suffering and developing a kind attitude to the self. Both MBSR and MBCL interventions will be taught by one of two accredited mindfulness teachers who have extensive experience in teaching MBIs, and who will complete the MBCL teaching training prior to the trial commencing. Adherence to the interventions will be measured by attendance at the group sessions and by participants home practice diaries. Fidelity to the interventions will be evaluated in line with guidance from previous studies and the application of a fidelity checklist.

Control condition: Prior to entering the intervention phase of the study, all individuals will begin in the control condition which consists of the routine medical monitoring and psychosocial support provided by gastroenterologists and IBD nurse specialists. Participants will be requested not to change their medication during the study, if at all possible, and to refrain from beginning any other psychological interventions.

Sample size: MBIs group sizes vary between 8 and 15 participants. Four groups will be conducted during the life of the grant, recruiting up to 60 participants. Despite being a pilot study we aim to achieve a sufficient sample size to adequately determine effectiveness. In line with previous studies of MBSR in chronic health conditions, assuming a conservative estimated medium effect size of d = .6 for our primary outcomes (e.g. depression and anxiety in diabetes) and a significance level of alpha = .05 (two-tailed), data from 45 participants would achieve 80% power45 and provide robust data for analysis.

Quantitative analysis: Statistical analysis will be carried out according to the principles of intention to treat. Repeated measures ANCOVAs will be conducted across all outcome measures, controlling for baseline measurements, to assess the potential impact of the intervention. Cohen's d effect sizes will be calculated to assess the magnitude of any potential change. In addition to the effectiveness of MBSR, and subsequently MBSR+MBCL, additional analyses to explore moderators of the treatment effects, such as disease type, age of diagnosis, current medication will be conducted. Sustainability of effects will be analysed via 3 and 6 month follow up data. The feasibility of the intervention will be evaluated via quantitative data on recruitment, enrolment, retention, attrition, missing data and fidelity to the model. Guidance on pilot and feasibility will be fully adhered to in reporting.

Qualitative Analysis: To assess the acceptability of the intervention, ascertain its value to participants and seek service-user views on any adaptations that would need to be made prior to a larger evaluation of the intervention, one-to-one interviews will be conducted with a sample of participants across the groups (aiming for a minimum of 12 participant interviews). All participants will be invited to take part, at the end of their respective group. The one-to-one interviews will be conducted by the lead researcher and be guided by an interview-schedule, designed to explore participants experience of the intervention in an open non-directive manner. Data will be transcribed and will be analysed using thematic analysis, which focuses on eliciting themes from participants' description of their experiences. Thematic analysis has been chosen as the methodology is not tied to a particular theoretical position, but offers a systematic approach to discerning themes in participant's accounts of their experiences.

Quality assurance plan: All aspects of the safety, monitoring and quality control of the data will be monitored by the a representative from the sponsor, there will be no separate Data Safety and Monitoring Board involved.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-25
* Confirmed diagnosis of IBD
* Be able to verbally communicate and write in English
* Be able to give informed consent
* Be able to engage in light exercise (required for the intervention)
* Be able to commit to home practice

Exclusion Criteria:

* Major psychiatric illness
* Active alcohol/drug dependency
* Scheduled for major surgery in the next 3 months
* Participation in any other IBD intervention studies within the last 6 months
* Prescribed antidepressants within the last 3 months.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Psychological Distress at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls.
  Psychological distress will be measured using 21-item The Depression Anxiety Stress Scales-Short Form (DASS-21). Participants will rate themselves on items such as, "I found myself feeling agitated, according to a 4-point Likert scale, higher scores indicating greater psychological distress. The measure yields three subscale scores: depression (range from 0 to 42), anxiety (range from 0 to 42), stress (range from 0 to 42), and an overall psychological distress total score (range from 0 to 126). The total score is computed by summing the subscale scores.
Change from Baseline Quality of Life at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Quality of life will be measured using the Inflammatory Bowel Disease Questionnaire (IBDQ). Participants rate themselves on items such as, "how frequent have your bowel movements been during the last two weeks?" according to seven point scales, lower scores indicating poorer health status in all subscales. The IBDQ is a 32-item self-report measure assessing quality of life, yielding four subscale scores: bowel symptoms (ranging from 10 to 70), systemic symptoms (range 5 to 35), emotional function (range 12 to 84) and social function (range 5 to 35) and a global subjective health status score calculated by summing the subscale scores (range from 32 to 224).
Change from Baseline Disease Activity at 3 time points | 8-weeks, 20 weeks, and 59 weeks.
  Disease activity will be measured by faecal calprotectin levels, a biological measure of disease activity. Calprotectin is activated when inflammation occurs (whatever the cause of that may be) and thus can be used as a diagnostic indicator. The concentration of calprotectin relates directly to the severity of the inflammation.

SECONDARY OUTCOMES:
Change from Baseline Mindfulness at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Mindfulness will be measured using the 15-item Five Facet Mindfulness Questionnaire. Participants will rate themselves on items such as, "When I'm walking, I deliberately notice the sensations in my body moving" according to a 5-point Likert scale, higher scores indicating greater mindfulness in all subscales. The measure yields five subscale scores: observing (range 8 to 40), describing (range 8 to 40), acting with awareness (range 8 to 40), non-judging of inner experience (range 8 to 40) and non-reactivity to inner experience (range 7 to 35) and a total score calculated by summing the subscale scores (range 39 to 195).
Change from Baseline Self-Compassion at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Self-compassion will be measured using the Self-Compassion Scale (SCS). Participants rate themselves on items such as, "I try to be loving towards myself when I'm feeling emotional pain" according to a 5-point Likert scale, higher scores representing greater self-compassion. The SCS yields six subscale scores: self-kindness (range 1 to 5), self-judgement (range 1 to 5), common humanity (range 1 to 5), isolation (range 1 to 5), mindfulness (range 1 to 5), overidentified (range 1 to 5) and a total score calculated by calculating a grand mean of the subscale means (range 1 to 5).
Change from Baseline Sleep Disturbance at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Sleep disturbance will be measured using the 8-item Patient-Reported Outcomes Measurement Information (PROMIS)-Sleep Disturbance Short-Form (SF) scale. Participants rate themselves on items such as, "My sleep was restless" according to a 5-point Likert scale, higher scores representing greater sleep disturbance. The PROMIS Sleep Disturbance measure yields one total score (range 8 to 40) calculated by summing the raw scores and converting them into a t-score.
Change from Baseline Fatigue at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Fatigue will be measured using the 8-item Patient-Reported Outcomes Measurement Information (PROMIS)-Fatigue Short-Form (SF) scale. Participants rate themselves on items such as, "I have trouble starting things because I am tired" according to a 5-point Likert scale, higher scores representing greater fatigue. The PROMIS Fatigue measure yields one total score (range 8 to 40) calculated by summing the raw scores and converting them into a t-score.
Change from Baseline Pain Interference and Intensity at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Pain Intensity and Interference will be measured using the 8-item Patient-Reported Outcomes Measurement Information (PROMIS)-Pain Interference Short-Form (SF) and the 1-item Patient-Reported Outcomes Measurement Information (PROMIS)-Pain Intensity Form. Participants will rate themselves on items such as, "How would you rate your pain on average?" according to a 7 and 5-point Likert scales respectively, higher scores representing greater pain interference and intensity. The PROMIS Pain Interference and Intensity measures yield two total scores (ranges 6 to 30 and 1 to 10 respectively) calculated by summing the raw scores and converting them into a t-scores.
Change from Baseline Coping Style at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Coping Style will be measured using the 28-item Brief Coping Orientation to Problems Experienced (COPE) measure. Participants will rate themselves on items about how often they had used different coping styles such as, "I've been saying to myself, this isn't real" according to a 4-point Likert scale, higher scores representing greater use of each coping style. The Brief COPE yield 14 subscales scores, of two items each (i.e., self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioural disengagement, venting, positive reframing, planning, humour, acceptance, religion and self-blame) calculated by summing the raw scores in each subscale (range 2 to 8 in all subscales).
Change from Baseline Self-Efficacy at 6 time points | When the intervention commences, 8-weeks, 12 weeks, 20 weeks, 33 weeks and 59 weeks; and at equivalent times for controls
  Self-efficacy will be measured using the 29-item Inflammatory Bowel Disease Self-Efficacy Scale (IBD-SES). Participants will rate themselves on items about how confident they feel in their ability to perform certain tasks such as, "Get emotional support from family and friends" according to a 10-point Likert scale, lower scores representing lower self-efficacy. The IBD-SES yields 4 subscales: managing stress and emotions (range 9-90), managing medical care (range 8 to 80), managing symptoms and disease (range 7 to 70), and maintaining remission (range 5 to 50) and a total score (range 29 to290) calculated by summing the raw scores in each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Rowse, Clin.Psy.D, Principal Investigator — University of Sheffield
Locations (1):
- Department of Clinical Psychology, University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan is to upload final anonymised data set to the Open Science Framework (OSF)
Supporting Information: Analytic Code
Time Frame: Data will become available when all analysis is complete and the findings are being prepared for publication
Access Criteria: Only the anonymised quantitative dataset will be made available
URL: https://osf.io/